CLINICAL TRIAL: NCT02880267
Title: Effectiveness and Safety of the Dexcom™ G6 Continuous Glucose Monitoring System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PTL-902220
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- CGM Users (Other): Glucose challenge during a clinic sessions to assess performance of CGM compared to reference measurement
  Interventions: Device: CGM

INTERVENTIONS:
Device: CGM — Glucose challenge during a clinic session to assess CGM performance compared to a laboratory reference measurement.

SUMMARY:
Effectiveness and Safety of the Dexcom G6 Continuous Glucose Monitoring (CGM) System

DETAILED DESCRIPTION:
The objective of the study is to establish performance of the System compared to a laboratory reference measurement. The effectiveness of the System will be evaluated by comparison of CGM values to a laboratory reference, Yellow Spring Instrument (YSI), using arterialized venous sample measurements. Performance will be evaluated in terms of point and rate accuracy of the System in reference to YSI.

The safety profile of the System will be characterized by the incidence of device-related Adverse Events (AEs) experienced by study subjects.

ELIGIBILITY:
Inclusion Criteria:

* Ages 2 or older
* Diagnosis of Type 1 diabetes or Type 2 diabetes, on intensive insulin therapy
* Willing to participate in a clinic session involving venous sampling for evaluation of study end point

Exclusion Criteria:

* Use of acetaminophen
* Known allergy to medical-grade adhesives
* Pregnancy
* Hematocrit outside specification of the study-assigned blood glucose meter

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Proportion of blood glucose values, compared between CGM and a lab glucose analyzer that are matched relative to a proportion of blood glucose values, compared between CGM and a lab glucose analyzer matched to an accuracy measurement of %20/20 mg/dL | 10 Days

CONTACTS AND LOCATIONS:
Overall Officials: David PRice, MD, Study Director — DexCom, Inc.
Locations (9):
- United States (9):
  - AMCR Institute, Escondido, California
  - Stanford, Palo Alto, California
  - Sansum, Santa Barbara, California
  - Diablo, Walnut Creek, California
  - Barbara Davis Center, Aurora, Colorado
  - Atlanta Diabetes, Atlanta, Georgia
  - Joslin Diabetes Center, Boston, Massachusetts
  - Oregon Health Science University, Portland, Oregon
  - Rainier, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No